CLINICAL TRIAL: NCT03594214
Title: Prognostic Value of Vitamin D Levels in Egyptian Females With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Barakat Saber, Principal investigator, Assiut University
Other Study IDs: Vitamin D in breast cancer
Record Dates: First submitted 2018-07-02; First posted 2018-07-20 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Vitamin D Deficiency
Keywords: breast cancer; vitamin d; prognosis
MeSH Terms: conditions — Vitamin D Deficiency; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: pre-treatment serum vitamin d level measured by ELISA kit in patients confirmed for diagnosis with invasive breast cancer and before receiving any treatment for breast cancer
  Interventions: Diagnostic Test: serum vitamin d level measured by ELISA kit

INTERVENTIONS:
Diagnostic Test: serum vitamin d level measured by ELISA kit — serum vitamin d level will be measured by a blood sample from newly diagnosed breast cancer patients just after diagnosis (either by surgery specimen or FNA or excisional biopsy specimen) and before receiving any type of treatment for breast cancer

SUMMARY:
In our study; we aim to analyze the correlation between pre-treatment serum vitamin D (VD) levels and breast cancer prognostic features in newly diagnosed breast cancer patients presenting to our department.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer diagnosed in females in more and less developed regions, with more cases occurring in less developed (883,000 cases) than more developed regions (794,000). In Egypt, breast cancer is the commonest cancer in females representing about (38.8%) of cancers in females.

Decades of epidemiologic research have led to the identification of a number of lifestyle and environmental breast cancer risk factors, including menstrual and/or reproductive history, use of hormones, anthropometry, and alcohol consumption, each typically explaining a modest proportion of the variation in disease risk.

Vitamin D exists as vitamin D2 (Calciferol, the storage form) and D3 (Cholecalciferol, the active form), which are metabolized to 25-hydroxyvitamin D [25(OH)D], the major circulating vitamin D metabolite; Besides, its physiological functions, vitamin D levels have also been studied as a risk factor for several hormonal cancers including breast cancer (BC). Vitamin D is not technically a vitamin, ie, it is not an essential dietary factor; rather, it is a pro-hormone produced photo-chemically in the skin from 7-dehydrocholesterol. The molecular structure of vitamin D is closely allied to that of classic steroid hormones (eg, estradiol, cortisol, and aldosterone) in that they have the same root ring structure. Technically, vitamin D is a secosteroid.

The vitamin D receptor (VDR) is a member of the nuclear receptor superfamily and plays a central role in the biological actions of vitamin D. The vitamin D receptor regulates the expression of numerous genes involved in calcium/phosphate homeostasis, cellular proliferation and differentiation, and immune response, largely in a ligand-dependent manner. To understand the global function of the vitamin D system in physio-pathological processes, great effort has been devoted to the detection of the vitamin D receptor in various tissues and cells, many of which have been identified as vitamin D targets.

According to a 2010 analysis, the vitamin D receptor significantly affects 229 human genes. Many of these genes have long been associated with autoimmune diseases and cancers. Greater than 36 types of tissue have been identified as having a Vitamin D Receptor including the breast .

In a study by. plasma vitamin D levels were correlated with deoxyribonucleic acid (DNA) repair capacity levels in women with breast cancer.

In another study there was an association between vitamin D insufficiency or deficiency and tumors with worse prognostic features. Low vitamin D levels were shown to be a risk factor for estrogen receptor (ER) negative tumors, with positive axilla and a higher rate of cell proliferation in Brazilian postmenopausal women.

A study that evaluated serum vitamin D levels in female patients with recently identified benign or malignant lesions of the breast and its associations with tumor histology. Vitamin D was associated with tumor aggressiveness.

However, the effect of vitamin D deficiency on breast cancer prognosis and its role as a non-invasive bio-marker of breast cancer outcomes warrants further investigation.

Newly diagnosed non-metastatic breast cancer patients presenting to clinical oncology department, Assiut university Hospitals will be assessed for pre-treatment serum vitamin D levels (classified as sufficiency (30-100 ng/mL), insufficiency (20- <30 ng/mL) and deficiency (<20 ng/mL) through a blood sample obtained from the patient before receiving any type of treatments for their cancer and analyzed using enzyme-linked immunosorbent assay (ELISA) kit for vitamin D serum levels, patients characteristics (age, menopausal status, body mass index (BMI as weight in kilograms divided by squared height in meters (kg/m2), data on breast cancer (histopathological type, grade, tumor stage, lymph node status), hormone status (estrogen receptor (ER), progesterone receptor(PR)), human epidermal growth factor receptor type 2 (HER2) and epithelial proliferative activity described in percentage (Ki-67) will be obtained from patient file records . Time to tumor relapse whether locally or distant metastases and overall survival will be recorded. Correlation between these data and the pre-treatment vitamin D levels will be done.

* Definition of menopause: the permanent cessation of menses for 12 consecutive months in the absence of chemotherapy, tamoxifen, toremifine, or ovarian suppression and follicle-stimulating hormone (FSH) and estradiol levels in the postmenopausal range.
* Tumor grade defined according to the Nottingham (also called Elston-Ellis) modification of the Scarff-Bloom-Richardson grading system Grade 1 tumor (well-differentiated). Grade 2 tumor (moderately differentiated). Grade 3 tumor (poorly differentiated).
* Tumor stage will be classified according to American Joint Committee on Cancer (AJCC) staging manual eighth edition (2017).
* Definition of HER-2 positivity according to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guideline recommendations for human epidermal growth factor receptor 2 (HER2) testing in breast cancer: Testing criteria define HER2-positive status when (on observing within an area of tumor that amounts to >10% of contiguous and homogeneous tumor cells) there is evidence of protein overexpression (IHC) or gene amplification (HER2 copy number or HER2/CEP17 ratio by ISH based on counting at least 20 cells within the area). If results are equivocal (revised criteria), reflex testing should be performed using an alternative assay (IHC or ISH).

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Newly diagnosed breast cancer patients.
* Histologically confirmed invasive breast carcinoma (IBC)
* Non- metastatic.
* Treatment naïve patients.
* Age: ≥18 and older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Patients must have normal organ function as regards LFTs and RFTs

Exclusion Criteria:

* Male patients
* Metastatic patients
* Previous history of breast cancer diagnosis or treatment
* Kidney impairment or renal stones
* History of parathyroidectomy
* Hypercalcemia, defined as serum level >11 mg/dl.
* Abnormal laboratory data for: AST (SGOT), ALT (SGPT), Serum Bilirubin, Alkaline phosphatase, Creatinine and/or Creatinine clearance, and Albumin.
* Female patients who are pregnant or breast feeding.
* Patients already on treatment or previously treated for vitamin D defeciency

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with newly diagnosed invasive breast cancer
Study Population: Female patients newly diagnosed with non-metastatic breast cancer, treatment-naive presenting to clinical oncology department at Assiut University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of vitamin D levels with prognostic features | 2 years
  Analysis of the correlation between; pre-treatment serum vitamin D levels, and breast cancer prognostic features.

SECONDARY OUTCOMES:
Correlation of vitamin d levels with treatment outcomes | 5 years
  Correlation between pre-treatment serum vitamin D levels, and disease free survival in years (DFS), overall survival in years (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Dina B Saber, Ass.Lecturer, Principal Investigator — Assiut University; Samir Sh Eid, professor, Study Director — Assiut University; Abeer F Amin, A.professor, Study Director — Assiut University; Maha S El-Naggar, lecturer, Study Director — Assiut University; Dalia T Kamal, lecturer, Study Chair — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Sousa Almeida-Filho B, De Luca Vespoli H, Pessoa EC, Machado M, Nahas-Neto J, Nahas EAP. Vitamin D deficiency is associated with poor breast cancer prognostic features in postmenopausal women. J Steroid Biochem Mol Biol. 2017 Nov;174:284-289. doi: 10.1016/j.jsbmb.2017.10.009. Epub 2017 Oct 12. PMID 29031688
- [Background] Ismail A, El-Awady R, Mohamed G, Hussein M, Ramadan SS. Prognostic Significance of Serum Vitamin D Levels in Egyptian Females with Breast Cancer. Asian Pac J Cancer Prev. 2018 Feb 26;19(2):571-576. doi: 10.22034/APJCP.2018.19.2.571. PMID 29481024